CLINICAL TRIAL: NCT04278001
Title: Clinical Usefullness of the Cuffless SOMNOtouch NIBP Device for 24-hour Ambulatory Blood Pressure Measurement
Acronym: BLAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Jakob Tobias Nyvad, Principal Investigator, Central Jutland Regional Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BLAST-AARHUS
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Arterial Hypertension
Keywords: Ambulatory blood pressure measurement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Masking Description: When evaluating data quality from either device, PI will be blinded to corresponding BP of the other device.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambulatory blood pressure measurement (Other): Dual 24-hour ABPM with both the SOMNOtouch NIBP and a validated oscillometric 24-hour ABPM-device (SPACELABS 90217 / 90207).
  Interventions: Device: Dual 24-hour ABPM

INTERVENTIONS:
Device: Dual 24-hour ABPM — Dual 24-hour ABPM with both the SOMNOtouch NIBP and a validated oscillometric 24-hour ABPM-device (SPACELABS 90217 / 90207).

SUMMARY:
The SOMNOtouch NIBP is a cuffless device for continuous blood pressure measurement. The device is widely used, but validation for 24-hour ambulatory blood pressure measurement (ABPM) is limited. This study seeks to validate the SOMNOtouch device for use in 24-hour ABMP as compared to a validated oscillometric device for 24-hour ABPM. A total of 60 patients with indication for 24-hour BP measurement will be recruited from our tertiary hypertension Clinic. All included patients will conduct dual 24-hour ABPM with both the SOMNOtouch NIBP and a the oscillometric device. Furthermore, patients will undergo measurement of arterial stiffness with a Sphygmocor device as well as complete a questionaire on device related discomfort.

DETAILED DESCRIPTION:
Recruitment of study participants:

A total of 60 patients with indication for 24-hour BP measurement will be recruited from our tertiary hypertension clinic at Aarhus University Hospital, Aarhus, Denmark. Patients will be eligible for inclusion if they are 18 years or older and have indication for ABPM with an automated oscillometric device. Exclusion criteria will be as follows: Known significant arterial abnormalities in the upper extremities, known cardiac arrythmia, upper arm circumference >16,5" or <6", or extreme uncontrolled hypertension (i.e. resting office BP > 230/140 mmHg). To enable testing of the device at both normal and elevated BP-levels, we will aim at including at least 15 patients in each of the following categories: Normal BP, stage 1 hypertension and stage ≥2, based on NICE guidelines for ABPM17. Informed consent will obtained from all patients prior to inclusion in the study. At inclusion, a simultaneous bilateral BP-measurement will be performed with three consecutive measurements using an automated oscillometric device (Microlife WatchBP Office®) after 5 minutes of rest. If the difference in Systolic Blood Pressure (SBP) between the arms is found to be >5 mmHg, the patient will not be included in the study.

24-hour BP measurements: All staff related to the project are familiar with the SOMNOtouch NIBP™ (SomBP) device, which has been used in our clinic for selected patients with high cuff-based BP and at the same time symptoms of hypotension, since 2015. Mounting and calibration of both devices will be conducted according to manufacturers' instructions. With the patient sitting in an upright position with back-support, a conventional oscillometric BP-device (Spacelabs 90217 / 90207, OscBP) will be fitted on the right arm, while the SomBP will be fitted on the left arm. The SomBP will be calibrated with a single BP measurement with a cuff-based sphygmomanometer. The OscBP will record BP three times every hour during daytime and two times every hour during nighttime, while the SomBP will measure BP continuously. The patients will be instructed to engage in normal activities but refrain from strenuous exercise and, at the time of cuff-inflation, to stop moving and talking, while keeping the arm still with the cuff at heart level. Pulse wave velocity (PWV) as well as pulse wave analysis (PWA) will be performed in duplicate with the SphygmoCor system (version 8.2, Atcor Medical, Sydney, Australia). A small questionnaire on device-related pain and/or discomfort as well as sleeping habits will be provided to all participants. As per ESH guidelines, a minimum of 70% useful measurements on the oscillometric device during the ABPM will be required for the data to be considered useful. Assessment the acceptability of data-quality of SomBP will be made on the basis of discussion between the primary investigator and KLC, who, at the time of evaluation will both be blinded to the corresponding OscBP measurement. No SomBP measurements will be accepted with more than 50% failed measurement in the report. Data from both devices will be excluded from the study if data-collection from either device is deemed to have insufficient quality to be usable. For these instances, patients will be asked to repeat examination with both devices. SomBP1 data will extracted ad hoc using Domino Light 1.4.0 software.

Statistical analysis:

All statistical analysis will be performed using STATA software. A p-value of 0.05 will be prespecified as statistically significant. Variables will be checked for distribution through histograms and QQ-plots. Means will be compared using paired t-test. Standard regression analysis will be performed to test for association in continuous variables. Categorical variables will be compared using chi-squared tests.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ABPM with an automated oscillometric device

Exclusion Criteria:

* Known significant arterial abnormalities in the upper extremities
* Known cardiac arrythmia
* Upper arm circumference >16,5" or <6", or
* Extreme uncontrolled hypertension (i.e. resting office BP > 230/140 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Difference in blood pressure averages between SOMNOtouch NIBP and SPACELABS 90217 / 90207 during 24-hour ABPM | During 24-hour ABPM
  in mmHg
Difference in mean systolic blood pressure between SOMNOtouch NIBP and SPACELABS 90217 / 90207 during 24-hour ABPM on the patient level | During 24-hour ABPM
  Bland Altman plots will be used to evaluate accuracy.
Difference in mean diastolic blood pressure between SOMNOtouch NIBP and SPACELABS 90217 / 90207 during 24-hour ABPM on the patient level | During 24-hour ABPM
  Bland Altman plots will be used to evaluate accuracy.

SECONDARY OUTCOMES:
The impact of aortic augmentation index normalized to a Heart frequency of 75 beats/minute on BP Measurements with either device. | Aortic augmentation index will be measured prior to 24-hour ABPM.
  As measured using the SphygmoCor-device
The impact of pulse wave velocity on BP Measurements with either device. | Pulse Wave velocity will be measured prior to 24-hour ABPM.
  As measured using the SphygmoCor-device
Patient satisfaction with SOMNOtouch device compared with the oscillometric device. | Immediately after completion om 24-hour ABPM.
  As judged based on standardized questionaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nyvad J, Christensen KL, Buus NH, Reinhard M. The cuffless SOMNOtouch NIBP device shows poor agreement with a validated oscillometric device during 24-h ambulatory blood pressure monitoring. J Clin Hypertens (Greenwich). 2021 Jan;23(1):61-70. doi: 10.1111/jch.14135. Epub 2020 Dec 17. PMID 33350030